CLINICAL TRIAL: NCT03358823
Title: Study on the Brain Network of Angelman Syndrome Based on Multi-modal Brain Image and Neural-EEG Data
Brief Title: Study on the Brain Network of Angelman Syndrome
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yi Wang, Vice Prsident Chlidren's Hospital of Fudan University, Fudan University
Other Study IDs: 2016YFC0904400
Record Dates: First submitted 2017-11-25; First posted 2017-12-02 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Angelman Syndrome
Keywords: AS database; MRI; EEG
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — whole blood 2*5ml, (isolate Plasma, Serum and white cell)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Angelman syndrome: Cases were children with the diagnosis meet the all 4 major criteria developmental delay, speech impairment, movement or balance disorder, and behavioral characteristics, as well as the presence of 3 of 6 minor criteria, including postnatal deceleration of head growth, seizures, abnormal EEG, sleep disturbance, attraction to or fascination with water, and drooling (summary by Tan et al., 2011). all patients meet the 4 known genetic mechanisms can cause Angelman syndrome (AS).,including maternal deletions involving chromosome 15q11.2-q13;paternal uniparental disomy of 15q11.2-q13;imprinting defectsand mutations in the gene encoding the ubiquitin-protein ligase E3A gene (UBE3A; 601623)

SUMMARY:
The aims of study on Angelman syndrome:

1. Establish the Angelman syndrome database
2. Explore the brain Network of Angelman Syndrome Based on Multi-modal Brain Image and Neural-EEG Data

DETAILED DESCRIPTION:
1. The participants recruitment: from Chinese Angelman Syndrome Patients group (Angelhome : angelman225@126.com) and Children's Hospital of Fudan University.
2. Fistly all participants had clinically and molecularly confirmed as Angelman syndrome . All participants should entry the online questionnaries and carified by telephone or on site . All the information will be recorded in the Angelman syndrome database. Investigators will analyze and summarize the relationship of phenotype and genotype(n=200).
3. Participants who assigned the informed consent and will undergo the brain MRI inspection and Neural-EEG recording in the Children's Hospital of Fudan University. The healthy age- and sex-matched control participants will enrolled in the same hospital. The Investigators will explore the brain morphology and electrophysiological alterations and for Angelman syndrome (AS) children among the different genotypes（n=200）.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and molecular diagnosis of Angelman syndrome.
* Agreed and completed the MRI scan and EEG-recording by using oral chloral hydrate.

Exclusion Criteria:

* Reject MRI scan and EEG-recording by using oral chloral hydrate or unable to complete the scan.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patients of Angelman syndrome meet the clinical and genetic diagnosis criteria
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Angelman syndrome databas; Brain Network of Angelman syndrome | 0-18 years old
  1. Analysis of geneal situation of Chinese Angelman syndrome including phenotype ,genotype, brain image ,EEG data, living quality ,comorbidy evolulation(n=200)
  2. Study on the Brain Network of Angelman Syndrome Based on Multi-modal Brain Image and Neural-EEG Data

CONTACTS AND LOCATIONS:
Overall Officials: Yi Wang, Dr., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghakhanyan G, Bonanni P, Randazzo G, Nappi S, Tessarotto F, De Martin L, Frijia F, De Marchi D, De Masi F, Kuppers B, Lombardo F, Caramella D, Montanaro D. From Cortical and Subcortical Grey Matter Abnormalities to Neurobehavioral Phenotype of Angelman Syndrome: A Voxel-Based Morphometry Study. PLoS One. 2016 Sep 14;11(9):e0162817. doi: 10.1371/journal.pone.0162817. eCollection 2016. PMID 27626634
- [Result] Tiwari VN, Jeong JW, Wilson BJ, Behen ME, Chugani HT, Sundaram SK. Relationship between aberrant brain connectivity and clinical features in Angelman Syndrome: a new method using tract based spatial statistics of DTI color-coded orientation maps. Neuroimage. 2012 Jan 2;59(1):349-55. doi: 10.1016/j.neuroimage.2011.07.067. Epub 2011 Jul 30. PMID 21827860